CLINICAL TRIAL: NCT06925646
Title: Hand Perfusion and Pulse Oximetry Performance
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Joyner, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 25-001363
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The study group will consist of 20 healthy non-smokers, with BMIs between 18-30 kg·m-2, free of cardiopulmonary diseases.
  Subjects will wear multiple pulse oximeter devices to measure arterial oxygen saturation (SpO2).
  Two fingers of each hand will be be equipped with identical FDA approved devices from two different commercial manufacturers.
  The third finger of each hand be equipped with a Mayo device developed by the SPPDG program for use by the US Military.
  Two wrist worn PPG-equipped "watches" (Garmin Fenix and the Mayo Clinic Developed SPPDG Watch) will be worn on each arm. One will be placed in the normal watch position (dorsal forearm) where pigmentation will generally be the darkest; the other will be placed on the volar forearm where pigmentation is generally less.
  Subjects will also have an indwelling catheter placed in the brachial artery to collect samples for blood gases.
  Interventions: Procedure: Finger hyperperfusion via adenosine; Procedure: Finger hypoperfusion via by norepinephrine; Procedure: Baseline hypoxic test

INTERVENTIONS:
Procedure: Finger hyperperfusion via adenosine — Subjects will be fitted with a mouthpiece and/or facemask to systematically reduce the fraction of inspired oxygen (FiO2) they breathe, starting with room air (21% O2), and then progressive hypoxic mixtures of 18%, 15%, 12%, and 10% FiO2 in sequence for five minutes each.
  Blood flow to the hand downstream from the brachial catheter will be increased by brachial artery infusions of adenosine administered at 6.25 mcg/100ml tissue per minute for 30 minutes into the brachial artery to increase blood flow by 5 to 10-fold.
Procedure: Finger hypoperfusion via by norepinephrine — Subjects will be fitted with a mouthpiece and/or facemask to systematically reduce the fraction of inspired oxygen (FiO2) they breathe, starting with room air (21% O2), and then progressive hypoxic mixtures of 18%, 15%, 12%, and 10% FiO2 in sequence for five minutes each.
  Blood flow to the hand downstream from the brachial catheter will be decreased to ~25% of baseline, by infusing norepinephrine at 4 ng/100ml of tissue per minute for 30 minutes.
Procedure: Baseline hypoxic test — Subjects will be fitted with a mouthpiece and/or facemask to systematically reduce the fraction of inspired oxygen (FiO2) they breathe, starting with room air (21% O2), and then progressive hypoxic mixtures of 18%, 15%, 12%, and 10% FiO2 in sequence for five minutes each.

SUMMARY:
The purpose of this study is to compare oxygen saturation measurement readings from manufactured pulse oximetry devices to the oxygen saturation measurements of arterial blood samples drawn at the same time of measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women of all races and ethnic backgrounds recruited from faculty and staff of the Mayo Medical Center and from Rochester, MN and surrounding communities.
* Equal number of male and female participants to address potential sex differences in physiology.
* We will intentionally recruit subjects with dark skin because of the issues surrounding accuracy of pulse oximetry and skin tone.
* Non-smokers
* BMIs between 18-30 kg·m-2.
* Female subjects will be non-pregnant.
* Free of cardiopulmonary diseases or other conditions and/or taking medications that might affect pulse oximeter-based estimates of arterial saturation.
* All inclusion and exclusion criteria are at the discretion of the Principal Investigator.
* At least 8 of the subjects will have Fitzpatrick Skin Type of IV to VI.

Exclusion Criteria:

• Children under the age of 18 will not be studied. We will exclude children less than 18 years of age because they are unable to give consent, and because these studies are non-therapeutic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of men and women of all races and ethnic backgrounds recruited from faculty and staff of the Mayo Medical Center and from Rochester, MN and surrounding communities.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygen saturation measured via arterial blood gas sample (Sa02) | 30 minutes, 90 minutes, 3 hours
  Arterial oxygen saturation will be obtained via a blood sample at the end of each stage of the breath down protocols and is reported as a percentage.
Arterial oxygen saturation measured via pulse oximeters (Sp02) | 30 minutes, 90 minutes, 3 hours
  Arterial oxygen saturation will be obtained via pulse oximeter reading at the end of each stage of the breath down protocols and is reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joyner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Department of Anesthesiology, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No